CLINICAL TRIAL: NCT00489645
Title: The Influence of Ambient Glycemia on the Effect of Pramlintide on Gastric Emptying in Patients With Type 1 Diabetes and Healthy Subjects
Brief Title: Effect of Hyperglycemia on Gastric Emptying Interactions With Pramlintide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: University of Rochester (Other)
Responsible Party: Joerg Schirra, MD, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: PRAM025/04; DFG Schi 527/1-2
Record Dates: First submitted 2007-06-19; First posted 2007-06-21 (Estimated); Last update posted 2008-01-16 (Estimated); Status verified 2008-01

CONDITIONS: Type 1 Diabetes
Keywords: pramlintide; gastric emptying; T1DM; postprandial
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — pramlintide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Placebo Comparator): Placebo, euglycemia
  Interventions: Drug: placebo
- 2 (Experimental): Pramlintide, euglycemia
  Interventions: Drug: pramlintide
- 3 (Placebo Comparator): placebo, hyperglycemia
  Interventions: Drug: placebo
- 4 (Experimental): pramlintide, hyperglycemia
  Interventions: Drug: pramlintide

INTERVENTIONS:
Drug: placebo — placebo SC during euglycemia
  Arms: 1
Drug: pramlintide — pramlintide SC during eglycemia
  Arms: 2
Drug: placebo — placebo during hyperglycemia
  Arms: 3
Drug: pramlintide — pramlintide SC during hyperglycemia
  Arms: 4

SUMMARY:
• To examine the influence of acute glycaemia (normoglycaemia and hyperglycaemia) on gastric emptying kinetics in patients with type 1 diabetes and non diabetic subjects when treated with subcutaneous (SC) injections of pramlintide.

DETAILED DESCRIPTION:
Postprandial increases in plasma glucose concentrations are mainly determined by the degree of postprandial suppression of endogenous glucose production and the rate of appearance of the ingested glucose. The latter is predominantly determined by the amount of glucose taken up by the splanchnic bed. Because nutrient absorption depends on gastric nutrient delivery, gastric emptying rate is a key determinant of the early rise of plasma glucose postprandially. At mealtime, the faster the stomach empties the more rapid the rise in plasma glucose. Yet, plasma glucose concentration is a determinant of gastric emptying rate. In non-diabetic subjects, as plasma glucose rises and approaches the upper limit of the normal range (~140 mg/dl), gastric emptying slows. This likely represents a physiological brake mechanism to limit excess delivery of nutrients, thus avoiding excessive appearance of glucose in plasma. In diabetes, abnormally accelerated gastric emptying as well as delayed gastric emptying have been reported. These conflicting data may be explained by differences of ambient glycaemia. In most of these studies undertaken in diabetic subjects these patients were severely hyperglycaemic, thus the reported delayed gastric emptying may be explained by the effect of hyperglycaemia on gastric motility. Indeed, a small number of studies controlled for ambient glycaemia found acceleration of gastric emptying in diabetes and suggest that diabetes manifests with a maladaptive acceleration of gastric emptying likely contributing to excessive postprandial plasma glucose excursions.

The amylin analog pramlintide is a potential new therapeutic that elicits a potent glucose lowering effect in the postprandial period thought to be due to both a suppression of plasma glucagon and a delay of gastric emptying. It is not clear, however, to what extent the pramlintide-induced delay of gastric emptying offsets a potential maladaptive acceleration of gastric emptying in diabetes patients studied under controlled glycemic conditions. In theory, every drug that reduces hyperglycaemia should accelerate gastric emptying and, thereby, minimize its potential effect on postprandial hyperglycaemia. Thus, the drug-induced effect of amylin on gastric motility may be of great advantage by offset the effects of glycemic induced acceleration on gastric emptying.

ELIGIBILITY:
Inclusion Criteria:

All of the following criteria are to be fulfilled for inclusion of an individual in the study unless the investigator grants an exception:

* Clinical diagnosis of type 1 diabetes (otherwise healthy) with an HbA1 ≤ 9%, and on a stable insulin treatment for at least 3 months (preferably on pump regimen) prior to screening OR is a healthy individual.
* 20-40 years of age, inclusive.
* Understand and sign an informed consent document, communicate with the investigator, and understand and comply with the requirements of the study.
* Euthyroid, including subjects receiving thyroid replacement therapy.

If female:

* Is surgically sterilized by hysterectomy; OR
* Is post-menopausal, as documented by a history of amenorrhea for 6 months and follicle stimulating hormone (FSH) level within the range specified as post-menopausal by the reporting laboratory at screen (post menopausal women on estrogen may enter the study without obtaining an FSH level); OR
* If of childbearing potential, meets the following criteria:

negative pregnancy test (ß-HCG), regardless of birth control method (including subjects with tubal ligation);

* Practicing and willing to continue throughout the study the appropriate contraception (defined as oral, injected, or implanted contraceptives for at least 3 months prior to entry, or barrier contraception).
* Agree to take every precaution to ensure that pregnancy will not occur during the study.

Exclusion Criteria:

* Individuals meeting any of the following criteria are to be excluded from the study unless the investigator grants an exception:
* History of severe hypoglycemia.
* Body mass index (BMI) ≥ 30 kg/m2.
* Autonomic nerve dysfunction: abnormal result in the cardiovascular parasympathetic and/or sympathetic tests (screening visit).

Hepatic disease:

* Known hepatic disease or transaminases (GOT, GPT) ≥ 2x above normal values.

Renal disease:

* Known or serum urea, serum creatinine ≥ 1.5x above normal values
* Cardiovascular or pulmonary disease:
* Arterial hypertension
* Blood pressure >150/95 mmHg at screening in a sitting position)
* Arterial occlusive disease
* Known coronary heart disease
* Abnormal ECG at screening visit.
* Gastrointestinal disease:
* Any known structural gastrointestinal disorder,
* Gastrointestinal surgery except for appendectomy,
* Symptoms indicating functional or structural upper gastrointestinal disorder (pain, bloating, postprandial fullness, nausea, emesis,
* Gastroectomy, gastroparesis, lactose intolerance, and diseases known to alter small bowel absorption; e.g., inflammatory bowel disease.

CNS disease:

* Epilepsy (including subjects with a past history of convulsions associated with hypoglycaemia),
* Psychiatric illness (including history of eating disorder such as bulimia or anorexia).
* Autoimmune disease other than thyroid, pernicious anemia, or vitiligo.
* Malignant disease requiring chemotherapy,
* Any acute febrile illness within 2 weeks of Screening (Visit 1) with a temperature of 100°F,
* Currently abusing alcohol or drugs, or have a history of alcohol or drug abuse that in the investigator's opinion could cause the subject to be non-compliant; or have a general history of non-compliance with medications.
* Receipt of any investigational drug within 90 days of Screening (Visit 1) (prior treatment with pramlintide is permissible).
* Currently treated with medications known to interfere with gastric emptying such as, but not limited to:

  * Ca2+ channel antagonists, ß-receptor antagonists, prokinetic agents metoclopramide (Reglan®) and cisapride (Propulsid®); and
  * Chronic (more than 10 days within a 6-month period) macrolide antibiotics such as erythromycin and newer derivatives.
* Currently treated with:

  * Bile acid sequestering resins cholestyramine (Questran®) and colestipol (Colestid®),
  * Systemic steroids,
  * Anti-obesity agents (including orlistat [Xenical®] and sibutramine [Meridia®]),
  * Alpha-glucosidase inhibitors (acarbose [Precose®] and miglitol [Glyset®]) and meglitinides ([Prandin®] and [Starlix®]).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2005-01; Primary Completion 2007-03 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
• To examine the influence of acute glycaemia (normoglycaemia and hyperglycaemia) on gastric emptying kinetics in patients with type 1 diabetes and non diabetic subjects when treated with subcutaneous (SC) injections of pramlintide. | 2 years

SECONDARY OUTCOMES:
• Gastric peristalsis derived from high-resolution scintigraphy by means of Fast Fourier Transform (FFT) analysis. • Effects on gastric emptying and on the rate of appearance of ingested glucose appearance, postprandial glucose sequestration, endoge | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Schirra, MD, Principal Investigator — Ludwig-Maximilians-University of Munic